CLINICAL TRIAL: NCT07201012
Title: Determining the Prevalence of Muir-Torre Syndrome in Patients With Lynch Syndrome
Acronym: SMT-SL
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIMAO/2024-01/EF-01
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Basal Cell Carcinoma of Skin, Site Unspecified; Epidermoid Carcinoma; Lynch Syndrome; Muir-Torre Syndrome
Keywords: Carcinoma; Screening; Skin cancer
MeSH Terms: conditions — Carcinoma, Basal Cell; Carcinoma, Squamous Cell; Colorectal Neoplasms, Hereditary Nonpolyposis; Muir-Torre Syndrome; Carcinoma; Skin Neoplasms

STUDY DESIGN:
Intervention Model Description: Sampling of suspected skin lesions (in accordance with good care practice) and swabbing of skin microbiota.
  Collection of previously excised cutaneous and deep tumour lesions kept in a public or private pathological anatomy facility for these patients.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Lynch syndrome undergoing screening for Muir-Torre syndrome (Other)
  Interventions: Diagnostic Test: Sampling of suspected skin lesions (in accordance with good care practices).; Genetic: Constitution of a biobank

INTERVENTIONS:
Diagnostic Test: Sampling of suspected skin lesions (in accordance with good care practices). — Sampling of suspected skin lesions (in accordance with good care practices) and swabbing of skin microbiota.
Genetic: Constitution of a biobank — Collection of previously excised cutaneous and deep tumour lesions kept in a public or private pathological anatomy facility for these patients

SUMMARY:
The main aim of this study is to determine the prevalence of Muir-Torre syndrome (MTS) in the population of patients with Lynch syndrome (LS) confirmed by genetic analysis. Other aims include describing the dermatological clinical manifestations of these patients in order to describe any possible new cutaneous manifestations of this syndrome. Another aim is to use molecular biology (microsatellite instability) and immunohistochemistry to analyze non-sebaceous skin lesions and deep-seated tumors that do not belong to the narrow spectrum of Lynch syndrome, and determine whether their occurrence in these patients is related to the genetic syndrome. The follow-up of these tumors (screening for new tumors) in patients with SL, as recommended by the learned societies, will also be evaluated. Finally, a biobank of cutaneous and deep tumour lesions in paraffin (retrospective) and smears of cutaneous lesions and healthy tissue (prospective) will be set up.

DETAILED DESCRIPTION:
Muir-Torre Syndrome (MTS) is an autosomal dominant disease described independently by Muir et al. in 1967 and Torre in 1968, defined by the association of a visceral tumor of the Lynch spectrum (colorectal, endometrial, urinary excretory tract, biliary tract, small intestine, stomach or glioblastoma carcinomas) and sebaceous skin tumors and/or multiple keratoacanthomas.

Histo-molecular examination of tumors for TMS/SL is based on 2 techniques, each focusing on a different aspect of TMS pathophysiology.

Immunohistochemistry (IHC) studies the presence of proteins from the MisMatch Repair (MMR) system in lesional tissues, and an absence of expression of one of these proteins is the physical translation of an abnormality in the MMR pathway, for which the presence of a constitutional mutation in one of the MMR system genes (MLH1, PMS2, MSH2, MSH6) is responsible. An IHC-deficient MMR phenotype (dMMR) results in a complete loss of expression of one or more MMR proteins in tumor cells, with expression maintained in "normal" cells (connective cells, immune cells, non-tumor epithelial cells).

Molecular biology or microsatellite instability (MSI) testing focuses on the molecular repercussions of MMR pathway failure. The aim of this technique is to determine the presence of microsatellite marker instability in tumor tissue. While for colorectal tumors, a comparative analysis of the patient's healthy tissue can be dispensed with, for other organs on the Lynch spectrum, including sebaceous tumors, a comparison with DNA from normal tissue can help interpret the results.

The incidence of TMS among patients with genetically proven SL is poorly known. Two studies have shown a prevalence of 9.2%, both involving American patients (1,2). These were 2 retrospective chart-based studies, the skin tumors not having been re-read for diagnostic confirmation.

These patients may also develop skin tumors not belonging to the SMT-SL spectrum, such as basal cell carcinomas (BCCs), squamous cell carcinomas (SCCs) or melanocytic tumors (melanomas and nevi). These skin and deep tumors (visceral tumors) not belonging to the Lynch spectrum of patients with proven SL have rarely been systematically studied for a dMMR phenotype.

French societies (INCa, Société Française de Gastroentérologie) have proposed the management of any patient with a mutation in one of the MMR system genes. Compliance with follow-up is a major public health issue. Digestive follow-up (regular colonoscopies) is only 68%, whereas gynecological follow-up is only 73% to 80%. Other types of follow-up, notably dermatological, have rarely been analyzed, and above all we have no data on compliance in France.

ELIGIBILITY:
Inclusion Criteria:

* Patient with a germline alteration of one of the MMR (MisMatch Repair) pathway genes (MLH1, PMS2, MSH2, MSH6) proven by constitutional genetic analysis (genetically authenticated Lynch syndrome).
* Patient followed at Nîmes University Hospital.
* Patient having given free and informed consent.
* Person affiliated to or benefiting from a social security scheme.

Exclusion Criteria:

* Person under court protection, guardianship or curatorship.
* A person who is unable to give consent.
* Person for whom it is impossible to give informed information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of Muir-Torre syndrome (MTS) in the population of patients with Lynch syndrome | Up to 6 months after inclusion
  Proportion of patients with Muir-Torre Syndrome confirmed by the occurrence of a sebaceous tumor (sebaceous adenoma, sebaceoma, sebaceous carcinoma) or several keratoacanthomas among patients with Lynch Syndrome. These tumors may or may not have had the mismatch repair system analyzed by immunohistochemistry (analysis of the 4 antibodies MLH1, PMS2, MSH2, MSH6) or by molecular biology (search for microsatellite instability).
  If the mismatch repair system has been studied, it must be deficient and the proteins absent on immunohistochemistry must be consistent with the mutated gene in Lynch Syndrome. If a block or slides are still available, sebaceous skin tumors or keratoacanthomas will be re-evaluated at Nîmes University Hospital for confirmation of the diagnosis.

SECONDARY OUTCOMES:
Dermatological clinical manifestations in patients with confirmed Lynch Syndrome | Up to 6 months after inclusion
  Presence of clinical dermatological signs associated with Lynch syndrome. YES/NO
Non-sebaceous skin lesions and Deep-seated tumors not belonging to the narrow spectrum of Lynch syndrome. Presence of antibody MLH1 | Up to 6 months after inclusion
  Molecular analysis (MSI test) and immunohistochemical analysis. Presence of antibody MLH1 on other tumour tissues (YES/NO) to determine the mismatch repair deficient (or MSI = pathological) or proficient (or MSS = normal) status of these lesions (and thereby their link with Muir-Torre syndrome).
Non-sebaceous skin lesions and Deep-seated tumors not belonging to the narrow spectrum of Lynch syndrome. Presence of antibody PMS2 | Up to 6 months after inclusion
  Molecular analysis (MSI test) and immunohistochemical analysis. Presence of antibody PMS2 on other tumour tissues (YES/NO) to determine the mismatch repair deficient (or MSI = pathological) or proficient (or MSS = normal) status of these lesions (and thereby their link with Muir-Torre syndrome).
Non-sebaceous skin lesions and Deep-seated tumors not belonging to the narrow spectrum of Lynch syndrome. Presence of antibody MSH2 | Up to 6 months after inclusion
  Molecular analysis (MSI test) and immunohistochemical analysis. Presence of antibody MSH2 on other tumour tissues (YES/NO) to determine the mismatch repair deficient (or MSI = pathological) or proficient (or MSS = normal) status of these lesions (and thereby their link with Muir-Torre syndrome).
Non-sebaceous skin lesions and Deep-seated tumors not belonging to the narrow spectrum of Lynch syndrome. Presence of antibody MSH6 | Up to 6 months after inclusion
  Molecular analysis (MSI test) and immunohistochemical analysis. Presence of antibody MSH6 (YES/NO) on other tumour tissues, to determine the mismatch repair deficient (or MSI = pathological) or proficient (or MSS = normal) status of these lesions (and thereby their link with Muir-Torre syndrome).

OTHER OUTCOMES:
Constitution of a biobank | Up to 6 months after inclusion
  Collection of previously excised cutaneous and deep tumour lesions kept in a public or private pathological anatomy facility for these patients

CONTACTS AND LOCATIONS:
Overall Officials: Pierre STOEBNER, Prof., Principal Investigator — Nîmes University Hospital

REFERENCES:
- [Background] Zhong CS, Horiguchi M, Uno H, Ukaegbu C, Chittenden A, LeBoeuf NR, Syngal S, Nambudiri VE, Yurgelun MB. Clinical factors associated with skin neoplasms in individuals with Lynch syndrome in a longitudinal observational cohort. J Am Acad Dermatol. 2023 Jun;88(6):1282-1290. doi: 10.1016/j.jaad.2023.01.035. Epub 2023 Feb 9. PMID 36773823
- [Background] South CD, Hampel H, Comeras I, Westman JA, Frankel WL, de la Chapelle A. The frequency of Muir-Torre syndrome among Lynch syndrome families. J Natl Cancer Inst. 2008 Feb 20;100(4):277-81. doi: 10.1093/jnci/djm291. Epub 2008 Feb 12. PMID 18270343
- [Background] Adan F, Crijns MB, Zandstra WSE, Bekkenk MW, Bleeker FE, Dekker E, van Leerdam ME. Cumulative risk of skin tumours in patients with Lynch syndrome. Br J Dermatol. 2018 Aug;179(2):522-523. doi: 10.1111/bjd.16552. Epub 2018 May 29. No abstract available. PMID 29542113
- [Background] Aziz S, O'Sullivan H, Heelan K, Alam A, McVeigh TP. Characterization of sebaceous and non-sebaceous cutaneous manifestations in patients with lynch syndrome: a systematic review. Fam Cancer. 2023 Apr;22(2):167-175. doi: 10.1007/s10689-022-00319-8. Epub 2022 Nov 23. PMID 36418753
- [Background] Latham A, Srinivasan P, Kemel Y, Shia J, Bandlamudi C, Mandelker D, Middha S, Hechtman J, Zehir A, Dubard-Gault M, Tran C, Stewart C, Sheehan M, Penson A, DeLair D, Yaeger R, Vijai J, Mukherjee S, Galle J, Dickson MA, Janjigian Y, O'Reilly EM, Segal N, Saltz LB, Reidy-Lagunes D, Varghese AM, Bajorin D, Carlo MI, Cadoo K, Walsh MF, Weiser M, Aguilar JG, Klimstra DS, Diaz LA Jr, Baselga J, Zhang L, Ladanyi M, Hyman DM, Solit DB, Robson ME, Taylor BS, Offit K, Berger MF, Stadler ZK. Microsatellite Instability Is Associated With the Presence of Lynch Syndrome Pan-Cancer. J Clin Oncol. 2019 Feb 1;37(4):286-295. doi: 10.1200/JCO.18.00283. Epub 2018 Oct 30. PMID 30376427
- [Background] Poumeaud F, Valentin T, Vande Perre P, Jaffrelot M, Bonnet D, Chibon F, Chevreau C, Selves J, Guimbaud R, Fares N. Special features of sarcomas developed in patients with Lynch syndrome: A systematic review. Crit Rev Oncol Hematol. 2023 Aug;188:104055. doi: 10.1016/j.critrevonc.2023.104055. Epub 2023 Jun 8. PMID 37301271